CLINICAL TRIAL: NCT02059161
Title: A Phase III Clinical Trial to Study the Safety and Efficacy of MK-1293 Compared to Lantus™ in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study of the Safety and Efficacy of MK-1293 Compared to Lantus™ in Participants With Type 1 Diabetes Mellitus (T1DM) (MK-1293-003)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1293-003; 2011-003971-12 (EudraCT Number)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — MK-1293; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-1293 (Experimental): MK-1293 dosed subcutaneously once daily at bedtime for 52 weeks. Doses were individually titrated post randomization to the suggested target for fasting fingerstick glucose levels of >70 mg/dL (3.9 mmol/L) and ≤100 mg/dL (5.6 mmol/L).
  Interventions: Drug: MK-1293; Drug: Prandial Insulin
- Lantus (Active Comparator): Lantus dosed subcutaneously once daily at bedtime for 52 weeks. Doses were individually titrated post-randomization to the suggested target for fasting fingerstick glucose levels of >70 mg/dL (3.9 mmol/L) and ≤100 mg/dL (5.6 mmol/L).
  Interventions: Drug: Lantus™; Drug: Prandial Insulin

INTERVENTIONS:
Drug: MK-1293 — MK-1293 dosed subcutaneously once daily at bedtime for 52 weeks. Initial dose will be determined based on the participant's previous insulin therapy. Thereafter, the dose will be titrated to the suggested target for fasting fingerstick glucose levels. MK-1293 dosing once daily at times other than bedtime will be permitted for participants with a previously established dosing time.
  Arms: MK-1293
Drug: Lantus™ — Lantus™ dosed subcutaneously once daily at bedtime for 52 weeks. Initial dose will be determined based on the participant's previous insulin therapy. Thereafter, the dose will be titrated to the suggested target for fasting fingerstick glucose levels. Lantus™ dosing once daily at times other than bedtime will be permitted for participants with a previously established dosing time.
  Other Names: Insulin glargine
  Arms: Lantus
Drug: Prandial Insulin — Participants will continue their prandial insulin during the study.

SUMMARY:
The purpose of this study is to compare the safety and efficacy of MK-1293 to Lantus™ in participants with T1DM. The primary hypothesis is that after 24 weeks, the mean change in hemoglobin A1c (A1C) from baseline is non-inferior in participants treated with MK-1293 compared with participants treated with Lantus™.

ELIGIBILITY:
Inclusion Criteria:

* T1DM For at least 1 year
* is currently using or has been using prandial insulin for at least 4 weeks. Participants taking any type of basal insulin should require a total daily dose of >=10 units/day. For participants currently taking pre-mixed insulin, the basal insulin component should be equivalent to a total daily dose of >=10 units/day.
* is male, or is female who is not of reproductive potential or if of reproductive potential agrees to remain abstinent or use (or have their partner use) an acceptable method of birth control during the study and for 14 days after the last dose of study medication

Exclusion Criteria:

* has had 1 or more severe hypoglycemic episodes associated with hypoglycemic seizure or loss of consciousness within the past 6 months
* history of ketoacidosis in the last 6 months
* participant, as assessed by the investigator, is not appropriate for or does not agree to target a fasting glucose of 70-100 mg/dL [3.9 -5.6 mmol/L].
* history of intolerance or hypersensitivity to Lantus™ or contraindication to Lantus™ or one of its excipients
* used a formulation of insulin glargine other than Lantus™
* has received injectable incretin-based therapy within the past 8 weeks
* on a weight loss program and not in the maintenance phase, or has started a weight loss medication within the past 8 weeks
* has undergone bariatric surgery within the past 12 months
* is likely to require treatment for 2 or more consecutive weeks or repeated courses of corticosteroids (note: inhaled, nasal, and topical corticosteroids are permitted)
* has undergone a surgical procedure within the past 4 weeks or has planned major surgery during the study
* has new or worsening signs or symptoms of coronary heart disease or congestive heart failure within the past 3 months, or has any following disorders within the past 3 months: acute coronary syndrome, coronary artery intervention, stroke or transient ischemic neurological disorder
* has severe peripheral vascular disease
* has high blood pressure
* has chronic myopathy, or a progressive neurological or neuromuscular disorder
* has active nephropathy
* history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* has human immunodeficiency virus (HIV)
* has a hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* history of malignancy in the past 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* history of melanoma, leukemia, lymphoma, or renal cell carcinoma
* is currently being treated for hyperthyroidism or has been on a stable dose of thyroid hormone replacement therapy for <6 weeks
* is a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence
* is pregnant or breast-feeding, or is expecting to conceive or donate eggs
* has donated blood products or has had phlebotomy of >300 mL within the past 8 weeks or intends to donate blood products during the study
* has poor mental function or works the night shift

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2015-05-04 (Actual); Study Completion 2015-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Home PD, Lam RLH, Carofano WL, Golm GT, Eldor R, Crutchlow MF, Marcos MC, Rosenstock J, Hollander PA, Gallwitz B. Efficacy and safety of MK-1293 insulin glargine compared with originator insulin glargine (Lantus) in type 1 diabetes: A randomized, open-label clinical trial. Diabetes Obes Metab. 2018 Sep;20(9):2220-2228. doi: 10.1111/dom.13354. Epub 2018 Jun 5. PMID 29766635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants at least 18 years of age who have had Type 1 diabetes mellitus (T1DM) for at least one year prior to study start.
Groups:
- MK-1293: MK-1293 dosed subcutaneously once daily at bedtime for 52 weeks. Doses were individually titrated post-randomization to the suggested target for fasting fingerstick glucose levels of >70 mg/dL (3.9 mmol/L) and ≤100 mg/dL (5.6 mmol/L).
Period: Overall Study
Arm/Group | MK-1293 | Lantus
Started | 245 | 263
Treated | 241 | 258
Completed | 196 | 222
Not Completed | 49 | 41
Not completed — Pregnancy | 0 | 2
Not completed — Adverse Event | 2 | 6
Not completed — Lost to Follow-up | 20 | 12
Not completed — Physician Decision | 4 | 4
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 16 | 13
Not completed — Randomized in error, no study drug | 0 | 1
Not completed — Non-compliance with study drug | 6 | 2

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1293 | Lantus | Total
Number analyzed (Participants) | 245 | 263 | 508
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (14.5) | 41.6 (14.8) | 41.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 111 | 217
  Male | 139 | 152 | 291

OUTCOME MEASURES:

1. Primary Outcome: Primary: Change From Baseline in Hemoglobin A1c (A1C) at Week 24
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). This change from baseline reflects the Week 24 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 24
Population: The analysis population included all randomized, treated participants who had at least one observation for the analysis endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
Percent | -0.62 [-0.79 to -0.45] | -0.66 [-0.82 to -0.50]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Non-Inferiority or Equivalence — The criterion for declaring non-inferiority was for the upper bound of the 95% CI to lie below 0.4%; Difference in the Least Squares Means = 0.04, 95% CI 2-sided [-0.11 to 0.19] — Longitudinal data analysis model included terms for treatment, time, prior insulin status (intermediate-acting, or long-acting insulin), and the interaction of time by treatment, and time by prior insulin status

2. Primary Outcome: Percentage of Participants With Any Confirmed Positive Anti-insulin Antibody (AIA) at Any Time Up Through Week 24
Description: Percentage of participants with confirmed positive AIA at any time up through Week 24 including baseline.
Time Frame: Up to Week 24
Population: The analysis population included all randomized, treated participants who had data for AIA at or before Week 24.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
Percentage of participants | 70.1 | 74.0
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Percentages = -3.9, 95% CI 2-sided [-11.8 to 4.0] — Miettinen & Nurminen

3. Primary Outcome: Percentage of Participants With Negative AIA at Baseline Who Develop Confirmed Positive AIA at Any Time Up Through Week 24
Description: Percentage of participants who became positive to AIA at or before Week 24, among participants who were AIA negative at baseline.
Time Frame: Up to Week 24
Population: The analysis population included all randomized, treated participants who were AIA negative at baseline and had data for AIA at or before Week 24.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 101 | 98
Percentage of participants | 32.7 | 35.7
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in Percentages = -3.0, 95% CI 2-sided [-16.1 to 10.1] — Miettinen & Nurminen

4. Primary Outcome: Change From Baseline in AIA Titer After 24 Weeks of Treatment
Description: This immunogenicity analysis will assess the effect of treatment with MK-1293 compared with Lantus on anti-insulin antibody development after 24 weeks of treatment. This change from baseline reflects the Week 24 AIA titer minus the Week 0 AIA titer.
Time Frame: Baseline and Week 24
Population: The analysis population included all randomized, treated participants who had AIA data at baseline and Week 24.
Measure: Mean (Standard Deviation); unit: AIA Titers
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 185 | 198
AIA Titers | 0.4 (15.9) | 0.3 (23.2)

5. Primary Outcome: Percentage of Participants Who Develop Insulin Neutralizing Antibodies Up Through Week 24
Description: Percentage of Participants Who Develop Insulin Neutralizing Antibodies Up Through Week 24. This immunogenicity analysis assessed the effect of treatment with MK-1293 and with Lantus on insulin-neutralizing antibody (INab) development up through 24 weeks of treatment.
Time Frame: Up to Week 24
Population: The analysis population included all randomized, treated participants who were INAb negative at baseline and who had data for INAb at or before Week 24.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 232 | 246
Percentage of participants | 3.9 | 5.3

6. Secondary Outcome: Change From Baseline in A1C at Week 52
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). This change from baseline reflects the Week 52 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
Percent | -0.35 [-0.53 to -0.17] | -0.33 [-0.50 to -0.16]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -0.02, 95% CI 2-sided [-0.18 to 0.14] — Longitudinal data analysis including terms for treatment, time, prior insulin status (intermediate-acting, or long-acting insulin), and the interaction of time by treatment, and time by prior insulin status

7. Secondary Outcome: Total Insulin Dose at Week 24
Description: Total insulin dose = basal insulin (MK-1293 or Lantus) + bolus (prandial) insulin (non-study medication).
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Insulin units
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 224 | 235
Insulin units | 58.74 [53.39 to 64.10] | 60.51 [55.21 to 65.81]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -1.77, 95% CI 2-sided [-4.69 to 1.16] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Total Insulin Dose Per Kilogram (kg) of Body Weight (Unit/kg) at Week 24
Description: Total insulin dose = basal insulin (MK-1293 or Lantus) + bolus (prandial) insulin (non-study medication).
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Insulin units/kg.
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 224 | 235
Insulin units/kg. | 0.75 [0.69 to 0.81] | 0.77 [0.72 to 0.83]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -0.02, 95% CI 2-sided [-0.06 to 0.01] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Blood glucose was measured on a fasting basis (collected after a 10-hour fast). FPG is expressed as mg/dL. This change from baseline reflects the FPG level at Week 24 minus the FPG level at Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
mg/dL | -16.8 [-33.4 to -0.2] | -26.4 [-42.5 to -10.3]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = 9.6, 95% CI 2-sided [-3.0 to 22.2] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Percentage of Participants With Confirmed Positive AIA Up Through Week 52
Description: Percentage of participants with confirmed positive AIA at any time up through Week 52 including baseline.
Time Frame: Up to Week 52 including baseline
Population: The analysis population included all randomized, treated participants who had data for AIA at or before Week 52.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
Percentage of participants | 73.4 | 75.6
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Differences in Percentages = -2.1, 95% CI 2-sided [-9.8 to 5.5] — Miettinen & Nurminen

11. Secondary Outcome: Percentage of Participants With Negative AIA at Baseline Who Develop Confirmed Positive AIA at Any Time Up Through Week 52
Description: Percentage of participants who became positive to AIA at or before Week 52, among participants who were AIA negative at baseline.
Time Frame: Up to Week 52
Population: The analysis population included all randomized, treated participants who had data for AIA at baseline and Week 52.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 101 | 98
Percentage of participants | 40.6 | 39.8
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in Percentages = 0.8, 95% CI 2-sided [-12.8 to 14.3] — Miettinen & Nurminen

12. Secondary Outcome: Change From Baseline in AIA Titer After 52 Weeks of Treatment
Description: This immunogenicity analysis assessed the effect of treatment with MK-1293 compared with Lantus on anti-insulin antibody development after 52 weeks of treatment. This change from baseline reflects the AIA titers at Week 52 minus the AIA titers at Week 0.
Time Frame: Baseline and Week 52
Population: The analysis population included all randomized, treated participants who had AIA data at baseline and Week 52.
Measure: Mean (Standard Deviation); unit: AIA Titers
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 164 | 177
AIA Titers | -1.6 (9.9) | 0.1 (20.3)

13. Secondary Outcome: Total Insulin Dose at Week 52
Description: Total insulin dose = basal insulin (MK-1293 or Lantus) + bolus (prandial) insulin (non-study medication).
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Insulin units
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 228 | 240
Insulin units | 59.16 [53.97 to 64.34] | 60.93 [55.79 to 66.06]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the least squares means = -1.77, 95% CI 2-sided [-4.92 to 1.39] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Total Insulin Dose Per Kilogram (kg) of Body Weight (Unit/kg) at Week 52
Description: Total insulin dose = basal insulin (MK-1293 or Lantus) + bolus (prandial) insulin (non-study medication).
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Insulin units/kg.
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 228 | 240
Insulin units/kg. | 0.75 [0.70 to 0.81] | 0.77 [0.71 to 0.82]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the least squares means = -0.02, 95% CI 2-sided [-0.05 to 0.02] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Change From Baseline in FPG at Week 52
Description: Blood glucose was measured on a fasting basis (collected after a 10-hour fast). This change from baseline reflects the FPG level at Week 52 minus the FPG level at Week 0.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
mg/dL | -17.9 [-35.8 to 0.1] | -12.5 [-29.9 to 4.9]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -5.4, 95% CI 2-sided [-19.7 to 8.9] — [estimate comment as in outcome 6, analysis 1]

16. Secondary Outcome: Percentage of Participants Who Develop Insulin Neutralizing Antibodies Up Through Week 52
Description: Percentage of Participants Who Develop Insulin Neutralizing Antibodies Up Thought Week 52. This immunogenicity analysis assessed the effect of treatment with MK-1293 and with Lantus on insulin-neutralizing antibody (INAb) development up through 52 weeks of treatment.
Time Frame: Up to Week 52
Population: The analysis population included all randomized, treated participants who were INAb negative at baseline and who had data for INAb at or before Week 52.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 232 | 246
Percentage of participants | 4.7 | 6.9

17. Secondary Outcome: Change From Baseline in 7-point Self-monitored Blood Glucose (SMBG) at Week 24
Description: The 7-point SMBG profile consisted of the following measurements by glucose meter: morning pre-meal (fasting), 2 hours after morning meal, midday pre-meal, 2 hours after midday meal, evening pre meal, pre-bedtime (pre-dose and at least 2 hours after evening meal), between 2:00 AM and 4:00 AM in the morning.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 226 | 248
mg/dL | -4.9 [-15.8 to 5.9] | -4.6 [-14.9 to 5.8]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -0.4, 95% CI 2-sided [-8.9 to 8.2] — Longitudinal data analysis model including terms for treatment, time, prior insulin status (intermediate-acting, or long-acting insulin), and the interaction of time by treatment, and time by prior insulin status

18. Secondary Outcome: Change From Baseline in 7-point SMBG at Week 52
Description: as for outcome 17
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 229 | 249
mg/dL | -12.0 [-25.8 to 1.7] | -4.0 [-16.3 to 8.4]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -8.1, 95% CI 2-sided [-18.6 to 2.4] — [estimate comment as in outcome 6, analysis 1]

19. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <7% and <6.5% After 24 Weeks of Treatment.
Description: Percentage of participants attaining A1C glycemic goals of <7.0% and <6.5% after 24 weeks of treatment.
Time Frame: 24 weeks
Population: The analysis population included all randomized, treated participants with a Week 24 A1C measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 219 | 236
Percentage of participants
  A1C < 7.0% | 37.0 | 37.7
  A1C < 6.5% | 20.5 | 21.6
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Adjusted Difference in %s (A1C < 7.0%) = -0.8, 95% CI 2-sided [-9.7 to 8.1] — Miettinen and Nurminen, stratified by prior insulin status
Statistical Analysis 2: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Adjusted Difference in %s (A1C <6.5%) = -1.1, 95% CI 2-sided [-8.6 to 6.5] — Miettinen and Nurminen, stratified by prior insulin status

20. Secondary Outcome: Percentage of Participants Attaining A1C Glycemic Goals of <7% and <6.5% After 52 Weeks of Treatment.
Description: Percentage of participants attaining A1C glycemic goals of <7.0% and <6.5% after 52 weeks of treatment.
Time Frame: 52 weeks
Population: The analysis population included all randomized, treated participants with a Week 52 A1C measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 197 | 221
Percentage of participants
  A1C < 7.0% | 31.0 | 30.8
  A1C < 6.5% | 14.2 | 18.6
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Adjusted Difference (A1C < 7.0%) = 0.2, 95% CI 2-sided [-8.7 to 9.1] — Miettinen and Nurminen
Statistical Analysis 2: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Adjusted Difference (A1C < 6.5%) = -4.4, 95% CI 2-sided [-11.5 to 2.8] — Miettinen and Nurminen

21. Secondary Outcome: Basal Insulin Dose at Week 52
Description: Basal Insulin Dose at Week 52.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
Units | 36.08 [33.14 to 39.03] | 36.51 [33.63 to 39.39]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in Least Means Squares = -0.42, 95% CI 2-sided [-2.33 to 1.48] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Basal Insulin Dose Per kg of Body Weight at Week 52
Description: Basal Insulin Dose per kg of Body Weight at Week 52.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units/kg
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
Units/kg | 0.46 [0.43 to 0.50] | 0.47 [0.43 to 0.50]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in Least Means Squares = -0.00, 95% CI 2-sided [-0.02 to 0.02] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Bolus Insulin Dose at Week 52
Description: Bolus Insulin Dose at Week 52.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 228 | 240
Units | 22.15 [19.03 to 25.27] | 23.65 [20.57 to 26.73]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -1.50, 95% CI 2-sided [-3.69 to 0.69] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Bolus Insulin Dose Per kg of Body Weight at Week 52
Description: Bolus Insulin Dose per kg of Body Weight at Week 52.
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units/kg
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 228 | 240
Units/kg | 0.28 [0.24 to 0.31] | 0.30 [0.26 to 0.33]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -0.02, 95% CI [-0.04 to 0.01] — [estimate comment as in outcome 1, analysis 1]

25. Secondary Outcome: Basal Insulin Dose at Week 24
Description: Basal Insulin Dose at Week 24.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
Units | 36.33 [33.24 to 39.42] | 37.07 [34.03 to 40.12]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -0.74, 95% CI 2-sided [-2.52 to 1.04] — [estimate comment as in outcome 1, analysis 1]

26. Secondary Outcome: Basal Insulin Dose Per kg of Body Weight at Week 24
Description: Basal Insulin Dose per kg of Body Weight at Week 24.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units/kg
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 241 | 258
Units/kg | 0.46 [0.43 to 0.50] | 0.48 [0.44 to 0.51]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -0.01, 95% CI 2-sided [-0.03 to 0.01] — [estimate comment as in outcome 1, analysis 1]

27. Secondary Outcome: Bolus Insulin Dose at Week 24
Description: Bolus Insulin Dose at Week 24.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 224 | 235
Units | 21.65 [18.50 to 24.81] | 22.91 [19.80 to 26.02]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -1.25, 95% CI 2-sided [-3.34 to 0.83] — [estimate comment as in outcome 1, analysis 1]

28. Secondary Outcome: Bolus Insulin Dose Per kg of Body Weight at Week 24
Description: Bolus Insulin Dose per kg of Body Weight at Week 24.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units/kg
Arm/Group | MK-1293 | Lantus
Number analyzed (Participants) | 224 | 235
Units/kg | 0.28 [0.24 to 0.31] | 0.29 [0.26 to 0.33]
Statistical Analysis 1: Comparison: MK-1293 vs Lantus; Test type: Superiority or Other; Difference in the Least Squares Means = -0.02, 95% CI 2-sided [-0.04 to 0.01] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: The safety population consisted of all randomized participants who received at least one dose of study treatment.
Arm/Group | MK-1293 | Lantus
Serious Adverse Events (participants affected / at risk) | 23/241 | 30/258
Other Adverse Events (participants affected / at risk) | 190/241 | 216/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1293 (N=241) | Lantus (N=258)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Oseomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (8) | 11 (14)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 2 (4) | 4 (4)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
VIth nerve paresis (Nervous system disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1293 (N=241) | Lantus (N=258)
Nasopharyngitis (Infections and infestations) | 19 (23) | 23 (29)
Upper respiratory tract infection (Infections and infestations) | 27 (40) | 28 (34)
Hypoglycaemia (Metabolism and nutrition disorders) | 185 (7617) | 204 (7544)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/ presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.